CLINICAL TRIAL: NCT04133207
Title: Registry Study of Patients With Advanced Breast Cancer Treated With Cyclin-dependent Kinase 4/6 (CDK4/6) Inhibitors Combined With Endocrine Therapy: the Experience of the Hellenic Cooperative Oncology Group
Brief Title: Clinical Outcome and Toxicity Data in Patients With Advanced Breast Cancer Treated With CDK Inhibitors Combined With Endocrine Therapy
Acronym: HeCOG/CDKi
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: CDK-HeCOG-2019
Record Dates: First submitted 2019-10-15; First posted 2019-10-21 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer Stage IV
Keywords: CDK; Breast cancer; toxicity; outcome
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from patients with breast cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with advanced HR-positive breast cancer: patients with histologically confirmed HR-positive, HER2-negative advanced (recurrent or metastatic) breast cancer. Patients had been treated in Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology

SUMMARY:
The present study will assess real-world clinical outcomes and adverse events from treatment with endocrine therapy combined with CDKi in patients with HR-positive, HER2-negative advanced breast cancer.

DETAILED DESCRIPTION:
Patients This will be a retrospective analysis of patients with histologically confirmed HR-positive, HER2-negative advanced (recurrent or metastatic) breast cancer. The investigators will use data from patients treated at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology. Eligible patients will be of 18 years or older, women of any menopausal status with HR-positive/HER2-negative advanced breast cancer who have received treatment with CDKi in combination with endocrine therapy for their advanced breast cancer. Treatment combinations of CDKi with any endocrine therapy will be accepted. Patients will be included in the analysis if they heve received at least two months of treatment with a CDKi. Patient clinical data will be obtained from their medical records. Toxicity data will be recorded from the clinicians' documentations during scheduled patient clinical visits.

Statistical analysis The primary endpoint of the study will be progression-free survival (PFS), defined as the time from treatment initiation to either the first documented disease progression or death from any cause. Secondary endpoint will be overall survival (OS), defined as the time from treatment initiation to patient death or last contact. Patients alive will be censored at the date of last contact. Adverse events will be graded based on Common Terminology Criteria for Adverse Events (CTCAE, version 4.0). Survival curves will be estimated using the Kaplan-Meier method and compared across groups with the log-rank test. The associations between the clinicopathological factors to be examined and the mortality rate will be evaluated with hazard ratios estimated with Cox proportional hazards model. The statistical analyses will be completed using the SAS software (SAS for Windows, version 9.3, SAS Institute Inc., Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Αny menopausal status is allowed
* HR-positive/HER2-negative advanced breast cancer
* Patients treated with CDKi in combination with endocrine therapy for their advanced breast cancer
* Combinations of CDKi with any endocrine therapy are allowed
* More than two months of treatment with a CDKi is mandatory

Exclusion criteria:

• Treatment with CDKi as (neo)adjuvant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective analysis of patients with histologically confirmed HR-positive, HER2-negative advanced (recurrent or metastatic) breast cancer. Patients had been treated in Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Toxicity rates | Time Frame: through the completion of the study, up to 2 years
  Rates of adverse events from the combination of CDKi and endocrine therapy

SECONDARY OUTCOMES:
Overall Survival | Time Frame: from the date of treatment start until death from any cause or date of last contact whichever occurred first, assessed up to 60 months
  Overall survival was defined as the time from diagnosis until death from any cause or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Oncology Cooperative Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fountzilas E, Koliou GA, Vozikis A, Rapti V, Nikolakopoulos A, Boutis A, Christopoulou A, Kontogiorgos I, Karageorgopoulou S, Lalla E, Tryfonopoulos D, Boukovinas I, Rapti C, Nikolaidi A, Karteri S, Moirogiorgou E, Binas I, Mauri D, Aravantinos G, Zagouri F, Saridaki Z, Psyrri A, Bafaloukos D, Koumarianou A, Res E, Linardou H, Mountzios G, Razis E, Fountzilas G, Koumakis G. Real-world clinical outcome and toxicity data and economic aspects in patients with advanced breast cancer treated with cyclin-dependent kinase 4/6 (CDK4/6) inhibitors combined with endocrine therapy: the experience of the Hellenic Cooperative Oncology Group. ESMO Open. 2020 Aug;5(4):e000774. doi: 10.1136/esmoopen-2020-000774. PMID 32817060